CLINICAL TRIAL: NCT01392859
Title: Characterization of the Role of Histamine in Children With Asthma
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Children's Mercy Hospital Kansas City (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: 105783-01
Record Dates: First submitted 2011-07-06; First posted 2011-07-13 (Estimated); Results first posted 2021-08-30 (Actual); Last update posted 2021-08-30 (Actual); Status verified 2021-08

CONDITIONS: Asthma; Allergic Asthma; Non-allergic Asthma
MeSH Terms: conditions — Asthma | interventions — levocetirizine; Solutions

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Initial Treatment: Levocetirizine(LCT) (Experimental): Group 1 will begin with active Levocetirizine(LCT) 0.5 mg/ml oral solution for 5-8 days. This arm will then undergo a 3-7 day washout period at which point crossover will occur and placebo will be provided for 5-8 days.
  Interventions: Drug: Levocetirizine 0.5 Mg/mL Oral Solution
- Initial Treatment: Placebo (Experimental): Group 2 will begin with placebo oral solution for 5-8 days. This arm will then undergo a 3-7 day washout period at which point crossover will occur and active Levocetirizine(LCT) 0.5 mg/ml will be provided for 5-8 days.
  Interventions: Drug: Levocetirizine 0.5 Mg/mL Oral Solution

INTERVENTIONS:
Drug: Levocetirizine 0.5 Mg/mL Oral Solution — Subjects in two arms, will be enrolled in a classical, randomized, double blind, crossover, placebo controlled trial of Levocetirizine(LCT) with determination of the PD response to LCT as determined by suppression of histamine microvasculature response via HILD.

SUMMARY:
Asthma, a chronic disease which produces significant morbidity and mortality in children, is a significant health problem to a large segment of society. Despite considerable advances in the diagnosis and treatment of asthma over the past several years, a sizeable portion of patients do not respond to the "core" treatments. The investigators are now learning that the underlying pathophysiology of disease is different among patients with asthma therefore; treatments which are beneficial in some patient groups may be not achieve affect in other groups.

Antihistamines have been studied in the past for the treatment of asthma. These studies have shown that there may be a beneficial effect of antihistamines in patients with allergic asthma where histamine likely plays a large role in disease and treatment response. However, there is not enough evidence to include these drugs in the standard treatment of asthma.

The investigators hypothesize that histamine plays a definable, significant role in disease pathogenesis and treatment response in children with allergic asthma. The investigators plan to test this overall hypothesis through two specific aims. The first aim will characterize the relative contribution of histamine in allergic vs. non-allergic asthma. This aim will be accomplished by comparison of the microvasculature response to histamine in children with allergic asthma and children with non-allergic asthma, measured by histamine iontophoresis with laser Doppler (HILD) monitoring, to determine potential phenotype-associated differences in the pharmacodynamic response to histamine.

ELIGIBILITY:
Inclusion Criteria:

* children age 7-17 years old
* with the diagnosis of allergic asthma or non-allergic asthma (n=102

Exclusion Criteria:

* history of immunodeficiency, mastocytosis
* chronic abnormal conditions of the skin, liver or kidney
* neoplastic disease
* movement or neurologic disorders
* active eczema on the forearms at the time of study
* history of a previous anaphylactic episode
* evidence of pregnancy (by urinary hCG) or lactation at the time of the study

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 211 (Actual)
Dates: Start 2011-06; Primary Completion 2015-03-29 (Actual); Study Completion 2015-03-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bridgette L. Jones, MD, Principal Investigator — Children's Mercy Hospital and Clinics
Locations (1):
- Children's Mercy Hospital and Clinics, Kansas City, Missouri, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 211 total participants enrolled in the study including the laser doppler testing. Only a small sub-set (n=28) of these participants were included in the sub-study including Levocetirizine.
Groups:
- Initial Treatment: Levocetirizine First, Then Placebo: Only a small sub-set of the overall study participants were included in this analysis.
  Group 1 will begin with active Levocetirizine(LCT) 0.5 mg/ml oral solution for 5-8 days. This arm will then undergo a 3-7 day washout period at which point crossover will occur and placebo will be provided for 5-8 days.
  These participants also went through the laser doppler portion prior to the crossover portion of the study.
  Levocetirizine 0.5 Mg/mL Oral Solution: Subjects in two arms, will be enrolled in a classical, randomized, double blind, crossover, placebo controlled trial of Levocetirizine(LCT) with determination of the PD response to LCT as determined by suppression of histamine microvasculature response via HILD.
- Initial Treatment: Placebo First, Then Levocetirizine: Only a small sub-set of the overall study participants were included in this analysis.
  Group 2 will begin with placebo oral solution for 5-8 days. This arm will then undergo a 3-7 day washout period at which point crossover will occur and active Levocetirizine(LCT) 0.5 mg/ml will be provided for 5-8 days.
  These participants also went through the laser doppler portion prior to the crossover portion of the study.
  Levocetirizine 0.5 Mg/mL Oral Solution: Subjects in two arms, will be enrolled in a classical, randomized, double blind, crossover, placebo controlled trial of Levocetirizine(LCT) with determination of the PD response to LCT as determined by suppression of histamine microvasculature response via HILD.
- Laser Doppler Portion Only: Participants who completed Only Laser Doppler portion of the study.
Period: Overall Study
Arm/Group | Initial Treatment: Levocetirizine First, Then Placebo | Initial Treatment: Placebo First, Then Levocetirizine | Laser Doppler Portion Only
Started | 15 | 13 | 183
Wash Out 3-7 Days | 15 | 13 | 0
Completed | 13 | 13 | 183
Not Completed | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall Study: 211 participants enrolled in overall study including laser doppler testing. Only 28 participants continued to subgroups below:
  Group 1: Initial Treatment: Levocetirizine(LCT) will begin with active Levocetirizine(LCT) 0.5 mg/ml oral solution for 5-8 days. This arm will then undergo a 3-7 day washout period at which point crossover will occur and placebo will be provided for 5-8 days.
  Levocetirizine 0.5 Mg/mL Oral Solution: Subjects in two arms, will be enrolled in a classical, randomized, double blind, crossover, placebo controlled trial of Levocetirizine(LCT) with determination of the PD response to LCT as determined by suppression of histamine microvasculature response via HILD.
  Group 2: Initial Treatment: Placebo will begin with placebo oral solution for 5-8 days. This arm will then undergo a 3-7 day washout period at which point crossover will occur and active Levocetirizine(LCT) 0.5 mg/ml will be provided for 5-8 days.
  Levocetirizine 0.5 Mg/mL Oral Solution: Subjects in two arms, will be enrolled in a classical, randomized, double blind, crossover, placebo controlled trial of Levocetirizine(LCT) with determination of the PD response to LCT as determined by suppression of histamine microvasculature response via HILD.
Arm/Group | Overall Study
Number analyzed (Participants) | 211
Age, Continuous [Mean (Standard Deviation); unit: Years] | 12.1 (3.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 90
  Male | 121
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 2
  Black or African American | 74
  White | 115
  More than one race | 17
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 211

OUTCOME MEASURES:

1. Primary Outcome: Characterize Contribution of Histamine in Children With Asthma
Description: The investigators will compare the response to histamine via histamine iontophoresis with laser doppler monitoring (measured in flux units on a continuous scale)between subjects with allergic asthma compared to subjects with non-allergic asthma.
Time Frame: one year
Population: Participants have been stratified based on their reactivity (i.e., participants with hyper-, normo-, or hypo-reactivity) and therefore the Number Analyzed for each Row differs from the Overall Number of Participants Analyzed.
Measure: Mean (Standard Deviation); unit: flux units on a continuous scale
Groups:
- Overall Study: Comparison of the microvasculature response to histamine in children with allergic asthma and children with non-allergic asthma, measured by histamine iontophoresis with laser Doppler (HILD) monitoring, to determine potential phenotype-associated differences in the pharmacodynamic response to histamine.
Arm/Group | Overall Study
Number analyzed (Participants) | 211
flux units on a continuous scale
  Hyper-Reactive-: number analyzed (Participants) | 83
  Hyper-Reactive- | 11253.24 (4271.17)
  Normo-Reactive: number analyzed (Participants) | 62
  Normo-Reactive | 6464.20 (1048.63)
  Hypo-Reactive: number analyzed (Participants) | 66
  Hypo-Reactive | 3539.67 (1239.95)

ADVERSE EVENTS:
Groups:
- Initial Treatment: Levocetirizine First, Then Placebo: Only a small sub-set of the overall study participants were included in this analysis.
  Group 1 will begin with active Levocetirizine(LCT) 0.5 mg/ml oral solution for 5-8 days. This arm will then undergo a 3-7 day washout period at which point crossover will occur and placebo will be provided for 5-8 days.
  Levocetirizine 0.5 Mg/mL Oral Solution: Subjects in two arms, will be enrolled in a classical, randomized, double blind, crossover, placebo controlled trial of Levocetirizine(LCT) with determination of the PD response to LCT as determined by suppression of histamine microvasculature response via HILD.
  These participants also went through the laser doppler portion prior to the crossover portion of the study.
  Note: Adverse Events (AE) were recorded by arm therefore AE's cannot be provided for each intervention separately. This data is no longer available to retrospectively separate AE's out by intervention.
- Initial Treatment: Placebo First, Then Levocetirizine: Only a small sub-set of the overall study participants were included in this analysis.
  Group 2 will begin with placebo oral solution for 5-8 days. This arm will then undergo a 3-7 day washout period at which point crossover will occur and active Levocetirizine(LCT) 0.5 mg/ml will be provided for 5-8 days.
  Levocetirizine 0.5 Mg/mL Oral Solution: Subjects in two arms, will be enrolled in a classical, randomized, double blind, crossover, placebo controlled trial of Levocetirizine(LCT) with determination of the PD response to LCT as determined by suppression of histamine microvasculature response via HILD.
  These participants also went through the laser doppler portion prior to the crossover portion of the study.
  Note: Adverse Events (AE) were recorded by arm therefore AE's cannot be provided for each intervention separately. This data is no longer available to retrospectively separate AE's out by intervention.
Arm/Group | Initial Treatment: Levocetirizine First, Then Placebo | Initial Treatment: Placebo First, Then Levocetirizine | Laser Doppler Portion Only
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/13 | 0/183
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/13 | 0/183
Other Adverse Events (participants affected / at risk) | 9/15 | 6/13 | 0/183
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Initial Treatment: Levocetirizine First, Then Placebo (N=15) | Initial Treatment: Placebo First, Then Levocetirizine (N=13) | Laser Doppler Portion Only (N=183)
Nausea (Gastrointestinal disorders) | 3 (3) | 2 (2) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0)
Chest Pain (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes